CLINICAL TRIAL: NCT02201043
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Phase II Clinical Study of Thalidomide in the Treatment of Ankylosing Spondylitis
Brief Title: Phase II Clinical Study of Thalidomide in the Treatment of Ankylosing Spondylitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Pharmaceuticals Holding Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SLDA-201
Record Dates: First submitted 2014-07-23; First posted 2014-07-25 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Ankylosing Spondylitis
Keywords: ankylosing spondylitis; thalidomide
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Thalidomide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Thalidomide 150mg (Active Comparator): Thalidomide 25mg/qd.po.2weeks; 50mg/qd.po.2weeks;100mg/qd.po.2weeks; 150mg/qd.po.to the end
  Interventions: Drug: Thalidomide 150mg
- Thalidomide 100mg (Active Comparator): Thalidomide 25mg/qd.po.2weeks; 50mg/qd.po.2weeks; 100mg/qd.po.to the end
  Interventions: Drug: Thalidomide 100mg
- Placebo (Placebo Comparator): Placebo po.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Thalidomide 150mg
  Other Names: Thalomid; Fan Ying Ting
  Arms: Thalidomide 150mg
Drug: Thalidomide 100mg
  Other Names: Thalomid; Fan Ying Ting
  Arms: Thalidomide 100mg
Drug: Placebo
  Arms: Placebo

SUMMARY:
1. Evaluate the efficacy and safety of taking thalidomide tablets once daily in the treatment of active ankylosing spondylitis.
2. To explore dose-effect relationships of taking thalidomide tablets once daily in the treatment of active ankylosing spondylitis, as well as selecting the appropriate dose for the further larger scale clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* (1) Active Ankylosing Spondylitis, Age 18-65, both outpatient or inpatient, both gender;
* (2) AS patients after traditional therapy (Using NSAIDs in a stable dose for 1 month, using oral corticosteroids, using NSAIDs for 3 months) still in active stage;
* (3) Pregnancy test must be negative in the female subjects of childbearing age or wife of the male subjects;
* (4)Female subjects with fertility during the trial (of 32 weeks) agreed to take a double medically accepted and reliable contraceptive measures, which includes a drug and a non-drug contraceptive measures; if the spouses of male subjects have fertility, agreed to use latex condoms for contraception;
* (5)Willing to have the treatment according to the plan as well as do the follow-up exam on time;
* (6)Understand and voluntarily signed informed consent.

Exclusion Criteria:

* (1) Suffering from or have suffered from rheumatoid arthritis, disc prolapse, septic arthritis, diffuse idiopathic skeletal hyperostosis syndrome, iliac dense osteitis, psoriatic arthritis, bowel disease arthritis, Reiter syndrome;
* (2) Severe AS, spine completely stiff (X-ray class IV) or the disease has been shown to have a shorter survival period;
* (3) Previously had total hip arthroplasty surgical treatment or appropriate to have the surgery;
* (4) Previously received anti-TNF therapy;
* (5) Used leflunomide within 3 months before screening;
* (6) Severe or persistent infection requires antimicrobial therapy;
* (7) Hepatitis B surface antigen or hepatitis C antibody test positive;
* (8) HIV positive or have acquired immunodeficiency syndrome (AIDS) history;
* (9) Malignancy, lymphoproliferative disease history;
* (10) Severe diabetes;
* (11) Resting hypotension (BP<90/50 mmHg) or hypertension (BP>170/100 mmHg), and orthostatic hypotension and clinically significant ECG abnormalities;
* (12) Over the past six months had a stroke, heart attack or other serious cardiovascular disease (including heart failure, unstable angina or life-threatening arrhythmias and coronary artery bypass graft surgery);
* (13) WBC or neutrophils below the lower limit of normal;
* (14) Liver dysfunction, AST or ALT l> 2 times the upper limit of normal;
* (15) Renal dysfunction, Cr>2 times the upper limit of normal;
* (16) Female subjects or spouses of male subjects have positive pregnancy test or be in the sickling period or intend to fertility or unwilling to take effective contraception;
* (17) With clinical symptoms of serious drug abuse or alcohol abuse or mental illness history;
* (18) Participated in any clinical trials of drugs within 3 months before screening;
* (19) Workers engaged in dangerous (eg drivers, machine operator, high-altitude operations, etc.);
* (20) A history of deep venous thrombosis or pulmonary embolism;
* (21) Be allergic to Test drug ingredients (including excipients);
* (22) Other reasons for not be enrolled.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2013-02; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Number of Subjects Achieving Assessment in Ankylosing Spondylitis 20 (ASAS 20) | week 12

SECONDARY OUTCOMES:
Change of ASDAS score | week 12
Change of ASDAS score | week 24
Mean change from baseline in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) | week 24
Mean change from baseline in Bath Ankylosing Spondylitis Function Index(BASFI) | week 24
Mean change from baseline in Nocturnal Pain using a Visual Analog Scale(VAS) | week 24
Mean change from baseline in back pain using a Visual Anolog Scale(VAS) | week 24
Morning stiffness | week 24
Number of Peripheral swollen joints | week 24
Number of Peripheral joint tenderness | week 24
Chest expansion | week 24
ESR | week 24
CRP | week 24
Schober test | week 24
Scoliosis | week 24

CONTACTS AND LOCATIONS:
Locations (9):
- China (9):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - The General Hospital of People's Liberation Army, Beijing, Beijing Municipality
  - Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Guanghua Hospital, Shanghai, Shanghai Municipality
  - Changhai Hospital, Shanghai, Shanghai Municipality
  - Xijing Hospital, XiAn, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - The Xinjiang Uygur Autonomous Region people's Hospital, Ürümqi, Xinjiang